CLINICAL TRIAL: NCT05249621
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of MZE001 to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Healthy Subjects
Brief Title: A Randomized Phase 1 of of MZE001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maze Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: MZE001-01
Record Dates: First submitted 2022-02-08; First posted 2022-02-21 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Mannitol; stearic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MZE001 (Experimental): MZE001 is a small molecule inhibitor of muscle glycogen synthase for the potential treatment of Pompe disease.
  Interventions: Drug: MZE001
- Placebo (Placebo Comparator): Excipients containing no active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MZE001 — Small molecule inhibitor of muscle glycogen synthase
  Other Names: MZ1449348
  Arms: MZE001
Drug: Placebo — Product containing excipients with no active ingredients
  Other Names: mannitol, silicified microcrystalline cellulose, magnesium stearate
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single (SAD) / multiple (MAD) ascending dose and food effect study.

DETAILED DESCRIPTION:
Phase 1 study is designed to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of orally administered MZE001 in healthy subjects, in fasted and fed states. Each SAD and MAD cohort will enroll 8 subjects randomized 6 active: 2 placebo to receive single or multiple doses of MZE001.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages 18 - 55 years, inclusive;
2. Must provide written informed consent prior to any study assessments and be willing and able to comply with all study procedures;
3. Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive;
4. Healthy as determined by the Investigator based on pre-study medical history, physical examination, and baseline safety laboratory studies.
5. Able to complete exercise treadmill test with no cardiac abnormalities detected
6. Females of childbearing potential who are sexually active with a non-sterilized partner must use a highly effective method of contraception during study participation and for 30 days after last administration of study drug.
7. Males of childbearing potential must use a highly effective method of birth control during study participation and for 90 days after last administration of study drug.

Exclusion Criteria:

1. Any concurrent condition that in the opinion of the Investigator would interfere with the evaluation of the investigational product or lead to increased risk of harm;
2. Any history of coronary artery disease or cardiovascular disease;
3. History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs;
4. History of cancer within past 5 years, with the exception of non-melanoma skin cancer and treated / excised melanoma;
5. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to the Screening visit;
6. Fridericia's corrected QT (QTcF) > 450 ms for male participants and > 470 ms for female participants or history of QT interval prolongation;
7. History or presence of an abnormal ECG that is clinically significant in the Investigator's opinion
8. Resting seated blood pressure < 90/40 mmHg or > 140/90 mmHg
9. Resting seated heart rate < 45 bpm or > 99 bpm
10. Poor peripheral venous access;
11. Have a history of drug hypersensitivity or anaphylaxis;
12. Current smoker or recent history of smoking within the last 3 months prior to the Screening visit;
13. Have a history of alcoholism or drug abuse or positive drug screen
14. Have used any prescription or non-prescription medicines or have been administered a vaccine within 14 days of admission,
15. Have received any investigational drug within 30 days or < 5 half-lives, whichever is longer, prior to the Screening visit;
16. Have donated or received any blood or blood products within the 3 months prior to the Screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of MZE001 | 14 days
  Occurrence of adverse events, serious adverse events, adverse events of special interest

SECONDARY OUTCOMES:
Maximum concentration following multiple doses of MZE001 | 14 days
  PK
AUC following multiple doses of MZE001 | 14 days
  PK
Accumulation ratio following multiple doses of MZE001 | 14 days
  PK

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Noonberg, MD, Study Director — Maze Therapeutics
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No